CLINICAL TRIAL: NCT06968403
Title: Community Emotional Intelligence Network to Address Mental Health Among Coastal Bangladeshis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Collaborators: Grand Challenges Canada (Other); Centre for Injury Prevention and Research Bangladesh (Other); University of Dhaka, Bangladesh (Other); North South University, Bangladesh (Unknown)
Responsible Party: Principal Investigator, Md Atiqul Haque, Professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1029; ST-POC-2312-62751 (Other Grant/Funding Number: Grand Challenges Canada)
Record Dates: First submitted 2025-04-30; First posted 2025-05-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Mental Health Conditions
Keywords: Emotional intelligence; Community mental health; Intervention; Bangladesh; coastal population

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volunteer and community participant (Experimental)
  Interventions: Behavioral: Community emotional intelligence network

INTERVENTIONS:
Behavioral: Community emotional intelligence network — This intervention focuses on developing emotional intelligence (EI) to tackle climate change-induced mental health challenges like eco-anxiety, solastalgia, and stress from displacement and natural disasters. It is community-centered, utilizing local resources and volunteers for EI training and mental health support, unlike traditional clinical interventions that depend on centralized healthcare systems. A mobile app is integrated to facilitate communication, learning resources, and participant connections, offering remote support and continuous engagement, even during climate events like floods or cyclones. Targeting coastal communities in Bangladesh, this program addresses the mental health impacts of frequent natural disasters, saltwater intrusion, and displacement. Unlike other mental health programs, it not only treats symptoms but also builds resilience against environmental stressors, empowering communities to cope with climate-induced mental health challenges.

SUMMARY:
The goal of this clinical trial is to learn if the community emotional intelligence network can improve mental health outcomes in coastal Bangladeshis affected by climate change and frequent natural disasters. The main questions it aims to answer are:

* Can enhancing emotional intelligence (e.g., self-awareness, empathy, emotional regulation, etc) improve the mental health of coastal Bangladeshis?
* Does the community emotional intelligence network increase resilience and coping strategies during climate-induced mental health crises? If there is a comparison group: NA

Participants will:

* Complete a pretested questionnaire focusing on socio-demographic characteristics, mental health impacts, and climate-change related stressors and perceptions
* Attend emotional intelligence training sessions focusing on self-awareness, self-regulation, empathy, and interpersonal skills
* Participate in follow-up assessments to evaluate mental health changes, emotional intelligence growth, and overall resilience
* Engage with a mobile app to facilitate communication, learning resources, and connection with other community members.

ELIGIBILITY:
Inclusion Criteria:

* - Aged 18 to 50 years
* Living in the selected study area for at least 6 months.
* Giving consent to participate in the intervention and follow-up.

Exclusion Criteria:

* Disability that hampers effective communication, either verbal or non-verbal.
* Undergoing end-stage illness depending on life-saving measures or palliative care.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Mental Well being | 8 weeks after completion of two-day intervention
  The WHO-5 Well-Being Index will be used to assess mental wellbeing both before and after the intervention. This tool consists of five statements, each rated on a Likert scale ranging from 'all of the time' to 'at no time'. Responses are scored on a scale from 0 to 5, with reverse scoring applied. Participants will evaluate each statement based on their experiences over the past two weeks. The total raw score, which ranges from 0 to 25, will then be multiplied by 4 to yield the final score, where a score of 0 represents the worst possible wellbeing and 100 represents the best. A raw score below 13 indicates poor wellbeing and serves as a potential indicator for depression.
Climate change related mental health status (Climate change anxiety scale) | 8 weeks after completion of two-day intervention
  Climate change-related mental health conditions of the participants will be measured by the Climate Change Anxiety Scale. It is a 22-item questionnaire on a Likert scale ranging from never to almost always. In this questionnaire, Items 1-13 constitute the climate change anxiety scale. Items 1-8 represent cognitive emotional impairment; 9-13 measure functional impairment; 14-16 measure experience of climate change; 17-22 measure behavioral engagement. This tool was culturally and linguistically validated before use. Proper permission was taken from the author for its use
Climate change related mental health status(Solastalgia scale;part of Environmental Distress Scale) | 8 weeks after completion of two-day intervention
  Solastalgia was measured using the Environmental Distress Scale. This scale has previously been used to measure the feelings of loss associated with solastalgia in the aftermath of specific events that caused environmental change or destruction. The EDS includes a sub-scale that measures solastalgia using ten items with possible scores ranging from 0-40. The solastalgia subscale has been used in prior research to assess solastalgia in the aftermath of environmental damage. This tool was culturally and linguistically validated before use. Proper permission was taken from the author for its use.
Mental Health (Depression, anxiety, stress) | 8 weeks after completion of two-day intervention
  The DASS-21 (Depression Anxiety Stress Scale - 21 items) is a self-report questionnaire designed to assess the severity of three related emotional states: depression, anxiety, and stress. It consists of 21 items, divided equally into three subscales, each containing 7 items. The depression subscale evaluates feelings of hopelessness and lack of interest, the anxiety subscale measures nervousness and physiological arousal, and the stress subscale gauges tension and irritability. Participants rate each item on a 4-point Likert scale (0-3), where higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Emotional Intelligence | 8 weeks after completion of two-day intervention
  Emotional intelligence of the participants will be assessed by the Trait Emotional Intelligence Questionnaire-Short Form (TEIQue-SF). This 30-item form includes two items from each of the 15 facets of the TEIQue. Items were selected primarily based on their correlations with the corresponding total facet scores, which ensured broad coverage of the sampling domain of the construct. The -SF can be used in research designs with limited experimental time or wherein trait EI is a peripheral variable. Although it is possible to derive from it scores on the four trait EI factors, in addition to the global score, these tend to have somewhat lower internal consistencies than in the full form of the inventory. The -SF does not yield scores on the 15 trait EI facets.

CONTACTS AND LOCATIONS:
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No